CLINICAL TRIAL: NCT00063284
Title: Safety Study of the Super Rapid Transcranial Magnetic Stimulation in Patients With Parkinson's Disease
Brief Title: Investigating the Safety of srTMS in the Treatment of Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030220; 03-N-0220
Record Dates: First submitted 2003-06-24; First posted 2003-06-25 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-04-15

CONDITIONS: Parkinson Disease
Keywords: Electrical Stimulation; Human Brain; Parkinson Disease; PD
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Device: Magstim Rapid Magnetic Stimulator

SUMMARY:
Super rapid transcranial magnetic stimulation (srTMS) is a method of brain stimulation that may be able to change the electrical activity of the nerve cells of the brain. It has been proposed and tested as a treatment for brain disorders, including Parkinson's disease.

The purpose of this study is to use a device called the magnetic stimulator to investigate the safe limit of srTMS, such as intensity of stimulation and the number of magnetic pulses that may lead to excessive brain stimulation.

Ten patients with Parkinson's disease-whose main problems are slowness of movement and difficulty walking-will participate in this study. They will be asked to come to the laboratory for one experiment. Before and after srTMS treatment, investigators will test participants' brain function with a series of psychological tests and an EEG (electroencephalogram). The srTMS treatment is performed by placing an insulated coil of wire on the scalp and passing a very brief electrical current through the wire coil. The experiment will last 2 to 4 hours.

DETAILED DESCRIPTION:
The treatment of Parkinson's disease (PD) needs further improvement, particularly in the areas of gait and freezing. A promising technique is repetitive transcranial magnetic stimulation (rTMS) that, so far, has produced small effects on bradykinesia in drug free patients in limited trials. The relevant rTMS parameters for the therapeutic effect are unknown. Use of very high rTMS frequency (50 Hz, maximum output of the modern TMS machines, super rapid TMS [srTMS] with circular coil design [vs. a figure eight shape]) may further improve the therapeutic effect in people who have PD. The 50 Hz srTMS frequency proposed here is in a range that exceeds the currently established guidelines since such high frequencies have not been investigated. We will look for acute srTMS effects of the primary motor cortex (M1) stimulation (60% to 100% motor threshold [MT] intensity, 0.5 seconds to 2 seconds train duration). A multi-channel electromyography (EMG) record will be visually controlled for signs of increasing time-locked EMG activity, EMG correlates of the spread of excitation through M1, or an increase of M1 excitability to establish the safe superrapid transcranial magnetic stimulation (srTMS) limit. The electroencephalogram (EEG) Record, Folstein Mini-Mental Exam, CFL and FAS Letter Production Test (words beginning with letters 'C', 'F' etc), Serial Reaction Time, Grooved Pegboard Test, and Unified PD Rating Scale (UPDRS) will be done before and after the srTMS session to control possible srTMS side effects.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects will be men and women aged 40 to 80 years with DOPA-responsive, akinetic-rigid PD.

After obtaining the informed consent, patients will be interviewed and examined by either the prinicipal investigator (PI) or a Brain Stimulation Unit (BSU) or an HMCS physician to establish the diagnosis of PD and rule out any other neurologic condition.

Only patients with a Hoehn and Yahr grade of 2 to 4 while 'off' will be accepted.

Patients must be on a regimen including L-DOPA, and they must have a total dose of medication equal to more than 300 mg of L-DOPA equivalent, including their dopamine agonist agents.

Any patient whose record does not contain a neurological examination from the past year will be reexamined before enrollment.

EXCLUSION CRITERIA:

Any significant medical or psychiatric illness (other than PD), pregnancy, history of epilepsy, or concurrent use of tricyclic antidepressants, neuroleptic agents, or any other licit or illicit drugs other than antiparkinsonian agents that could lower the seizure threshold.

Persons with surgically or traumatically implanted foreign bodies such as a pacemaker, or any implanted stimulators, an implanted medication pump, a metal plate in the skull, or metal inside the skull or eyes (other than dental appliances or fillings) that may pose a physical hazard during magnetic stimulation will also be excluded.

Most of these exclusions also come under the category of significant medical illness. Patients for whom participation in the study would, in the opinion of the investigators, cause undue risk or stress for reasons such as tendency to fall, excessive fatigue, general fatigue, general frailty, or excessive apprehensiveness will also be excluded.

A urine sample for the pregnancy test will be obtained from any women of childbearing potential prior to the start of srTMS, on the day of the initial interview and signing of the consent form. Pregnant women will be excluded from the study.

Mentally impaired patients who have no capacity to provide their own consent will be excluded from the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2003-06-18; Study Completion 2009-04-15

PRIMARY OUTCOMES:
Testing the safety limit (SL) of 50 Hz srTMS. | Single visit

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Baudewig J, Siebner HR, Bestmann S, Tergau F, Tings T, Paulus W, Frahm J. Functional MRI of cortical activations induced by transcranial magnetic stimulation (TMS). Neuroreport. 2001 Nov 16;12(16):3543-8. doi: 10.1097/00001756-200111160-00034. PMID 11733708
- [Background] Aarsland D, Larsen JP, Waage O, Langeveld JH. Maintenance electroconvulsive therapy for Parkinson's disease. Convuls Ther. 1997 Dec;13(4):274-7. PMID 9437571
- [Background] Belmaker RH, Grisaru N. Magnetic stimulation of the brain in animal depression models responsive to ECS. J ECT. 1998 Sep;14(3):194-205. PMID 9773358